CLINICAL TRIAL: NCT05594979
Title: An Open-label, Single Center, Single Arm, Clinical Trial to Assess the Consumption Effects of 6 Weeks TOTUM-070 on Lipid Metabolism and Cardiovascular Health in Individuals at Increased Cardio-metabolic Risk
Brief Title: Effects of 6 Weeks TOTUM-070 on Lipid Metabolism and Cardiovascular Health in Individuals at Increased Cardio-metabolic Risk
Acronym: OLALIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment period has come to an end and will not be renewed due to insufficient recruitment.
Sponsor: Valbiotis (Industry)
Collaborators: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VCT-015; 2022-A01474-39 (Other: ID-RCB)
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Hypercholesterolemia; Cardiovascular Risk Factor; Dyslipidemias; Atherosclerosis; Cardio-metabolic Risk
Keywords: Moderate hypercholesterolemia; Nutrition healthcare; Plant extracts
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOTUM-070 (Experimental): Experimental active diet supplement TOTUM-070 taken 2 times per day
  Interventions: Dietary Supplement: TOTUM-070

INTERVENTIONS:
Dietary Supplement: TOTUM-070 — 2.5-g dose of TOTUM-070 diet supplement; Four capsules per day to consume orally in two intakes

SUMMARY:
This clinical study aims to assess the efficacy of 6 weeks 2.5g dose of TOTUM-070, a mix of 5 plant extracts, on lipid metabolism and cardiovascular health in individuals at increased cardio-metabolic risk.

ELIGIBILITY:
Main Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 35 kg/m²
* Moderate hypercholesterolemic subject without any clinical symptoms of hypercholesterolemia (xanthoma, recurrent chest and/or leg pain…) and not requiring immediate pharmacological lipid-lowering treatment according to the current recommendations (European Society of Cardiology /European Atherosclerosis Society, 2019)
* Fasting blood LDL cholesterol level (using Friedewald estimation method) between 1.3 and 1.9 g/L
* Fasting blood triglycerides level ≤ 2.2 g/L

Main Exclusion Criteria:

* Suffering from a metabolic disorder such as diabetes, uncontrolled thyroidal dysfunction or other metabolic disorder needing a dose adjustment in drug intervention according to the professional recommendations
* Suffering from an uncontrolled arterial hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg)
* With a history of ischemic cardiovascular event
* Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, ongoing hepatic or biliary disorders, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease)
* Fasting glucose plasma concentration > 1.26 g/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline of blood LDL cholesterol concentration at 6 weeks | V1 (baseline) and V2 (6 weeks of intervention)
  LDL cholesterol (Friedewald method)

SECONDARY OUTCOMES:
Change from baseline of the fasting blood concentration of triglycerides | V1 (baseline) and V2 (6 weeks of intervention)
  Triglycerides
Change from baseline of the fasting blood concentration of total cholesterol | V1 (baseline) and V2 (6 weeks of intervention)
  Total cholesterol
Change from baseline of the fasting blood concentration of HDL cholesterol | V1 (baseline) and V2 (6 weeks of intervention)
  HDL cholesterol
Change from baseline of the fasting blood concentration of non-HDL cholesterol | V1 (baseline) and V2 (6 weeks of intervention)
  Non-HDL cholesterol
Change from baseline of the fasting blood concentration of free fatty acids | V1 (baseline) and V2 (6 weeks of intervention)
  Free fatty acids
Change from baseline of the fasting blood concentration of apolipoprotein-A1 | V1 (baseline) and V2 (6 weeks of intervention)
  Apolipoprotein-A1
Change from baseline of the fasting blood concentration of apolipoprotein-B | V1 (baseline) and V2 (6 weeks of intervention)
  Apolipoprotein-B

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Clermont Ferrand, Clermont-Ferrand, France